CLINICAL TRIAL: NCT02977403
Title: Pilot Study of Mobile Attention Training in Overweight Female Adolescents
Brief Title: Mobile Attention Retraining in Overweight Female Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 170014; 17-CH-0014 (Other: NIH Clinical Center)
Record Dates: First submitted 2016-11-29; First posted 2016-11-30 (Estimated); Results first posted 2024-08-20 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Overweight; Binge Eating; Healthy Volunteers
Keywords: Binge Eating; Eating Behavior; Children; Magnetoencephalography; Loss of Control
MeSH Terms: conditions — Obesity; Overweight; Bulimia; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Overweight youth with loss of control over eating randomized to intervention or control groups Overweight youth without loss of control over eating randomized to intervention or control groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Assignment to intervention or control made by a person who has no contact with study subjects to place the appropriate program on the phone used by the subject. Blind was maintained until all subjects had completed all assessments for the randomized phase.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB Retraining (Experimental): Active treatment - the probe always replaces the neutral picture. There is a perfect correlation between picture type and probe location.
  Interventions: Behavioral: Attention Bias Retraining
- Control sham (Sham Comparator): Sham Comparator program - the probe randomly replaces the neutral or food picture. There is no correlation between picture type and probe location
  Interventions: Behavioral: Sham Comparator: AB Control

INTERVENTIONS:
Behavioral: Attention Bias Retraining — Attention retraining program on smartphone where the probe always replaces the neutral picture. There is a perfect correlation between picture type and probe location.
  Arms: AB Retraining
Behavioral: Sham Comparator: AB Control — Sham Comparator "training" where the probe randomly replaces the neutral or food pictures. There is no correlation between picture type and probe location
  Arms: Control sham

SUMMARY:
Background:

People are constantly exposed to unhealthy foods. Some studies of adults show that training attention away from unhealthy foods might reduce overeating. Researchers want to see what happens in the brain when teens train their attention away from food through a program on a smartphone.

Objective:

To study the relationship between eating patterns, body weight, and how the brain reacts to different images.

Eligibility:

Right-handed females ages 12-17 who are overweight (Body Mass Index at or above the 85th percentile for age).

Design:

Participants will have 6 visits over about 8 months.

Visit 1: participants will be screened with:

Height, weight, blood pressure, and waist size measurements

Medical history

Physical exam

Urine sample

DXA scan. Participants will lie on a table while a very small dose of x-rays passes through the body.

Questions about their general health, social and psychological functioning, and eating habits

Parents or guardians of minor participants will answer questions about their child s functioning and demographic data.

Before visits 2-6, participants will not eat or drink for about 12 hours. These visits will include some or all of these procedures:

Blood drawn

MRI scan. Participants will lie on a stretcher that slides in and out of a metal cylinder in a strong magnetic field. A device will be placed over the head.

Meals provided. Participants will fill out rating forms.

Simple thinking tasks

A cone containing magnetic field detectors placed onto the head

Medical history

Physical exam

Urine sample

Participants will be assigned to a 2-week smartphone program that involves looking at pictures. Participants will complete short tasks and answer some questions about their eating habits and mood on the smartphone.

DETAILED DESCRIPTION:
Over 30% of adolescents are overweight and 20% are obese, but the mechanisms that produce excessive weight gain in youth remain incompletely elucidated. Some overweight youth appear to have an attention bias (AB: a tendency to attend selectively to stimuli that have acquired salience or meaning) toward highly palatable food that may lead to overeating. AB involves distinct cognitive processes, (1) unconscious reactions (UCR), reflecting initial attention capture evoked by salient stimuli, and (2) continued attention deployment (AD) to stimuli relevant to current goals. These rapidly evolving processes are associated with unique neurocircuitry best measured using high spatial resolution and temporal sensitivity. Magnetoencephalography (MEG) is a novel neuroimaging technology that has both excellent temporal and good spatial resolution, thus is uniquely and ideally suited to study neurocognitive mechanisms of AB. Reducing AB to palatable foods may help some overweight youth curb their consumption of energy-dense options. Attention retraining (AR) programs can be used to reduce AB and have been effective in reducing AB to unhealthy food in adults. Although most AR studies involve computers in the laboratory, using smartphones in the natural environment may be a particularly effective method to deliver AR to adolescents and measure AB using ecological momentary assessment. The first aim of the proposed study is to investigate, using MEG, the impact of a 2-week smartphone AR program on neural responses to food cues in overweight adolescent (12-17 y/o) girls with and without loss of control (LOC) eating, defined as a subjective experience of a lack of control over what or how much one is eating. LOC is a distinct eating behavior phenotype in youth that is a risk factor for excess weight gain and disordered eating, and is much more prevalent among girls (vs. boys). Overweight youth who report LOC may be particularly susceptible to AB. Additionally, adults with LOC demonstrate AB toward socially threatening cues, such as angry or disapproving faces, and the AB to social threat may be relevant to the relationship between AB to food and overweight. The second goal is to examine the effect of the 2-week AR program on AB, food intake, and body composition. An exploratory aim is to examine whether AB to socially threatening cues, moderates the effects of this novel intervention on AB to food cues, food intake, and body composition. The proposed study is innovative because no study to date has examined neurocircuitry of ABs to food using MEG, nor examined the impact of AR delivered in the natural environment on neurocircuitry of AB in a group of youth prone to AB. These studies may help further characterize phenomenology of distinct obesity subtypes and may potentially identify an approach that could prevent undue weight gain in adolescent girls at risk for obesity.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers will qualify if they meet the following criteria:

1. Age between 12 and 17 years (at the start of the study).
2. Female sex.
3. BMI at or above the 85th percentile for age and sex according to the Centers for Disease Control US Standards (101).
4. Right handedness.

   LOC sample only:
5. Greater than or equal to 1 episodes of LOC eating during the past month prior to assessment, assessed using a clinical diagnostic interview for eating disorders.

   No-LOC sample only:
6. No episodes of LOC eating during the past month prior to assessment, assessed using a clinical diagnostic interview for eating disorders.

EXCLUSION CRITERIA:

Individuals will be excluded (and provided treatment referrals as needed) for the following reasons:

1. An obesity-related health comorbidity requiring medical treatment, such as hypertension (defined by age-, sex-, and height-specific standards) or fasting hyperglycemia consistent with diabetes.
2. Presence of other major illnesses: renal, hepatic, gastrointestinal, most endocrinologic (e.g., Cushing syndrome, untreated hyper- or hypothyroidism), hematological problems or pulmonary disorders (other than asthma not requiring continuous medication). Nonserious

   medical illnesses, such as seasonal allergies, will be reviewed on a case-by-case basis.
3. Regular use of any medication known to affect body weight or eating behavior (e.g., stimulants prescribed for attention deficit hyperactivity disorder, or ADHD). Medication use for non-serious conditions (e.g., acne) will be considered on a case-by-case basis.
4. Current pregnancy or a history of pregnancy.
5. A significant reduction in weight during the past three months, for any reason, exceeding 5% of body weight.
6. Presence in the child of any significant, full-threshold psychiatric disorder based on DSM criteria (102), such as schizophrenia, bipolar disorder, alcohol or substance abuse, anorexia or bulimia nervosa, or any other disorder that, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study. These individuals will not be permitted to enroll in the current study and will be referred for treatment. Individuals who present with other psychiatric disorders, including subthreshold psychiatric disorders, will be permitted to enroll in the study. If, based on the opinion of the investigators, a participant requires treatment for his/her psychiatric symptoms, the individual will be referred for treatment. Participants who develop any psychiatric disorder or significant psychiatric symptoms at any follow-up assessment during the study will be excluded and be provided with treatment referrals.
7. Current and regular substance use, including the use of alcohol and/or tobacco products (including e-cigarettes).
8. A history of significant or recent brain injury that may considerably influence performance (i.e., any history of loss of consciousness greater than or equal to 30 minutes associated with a head injury, any history of memory loss or hospitalization associated with a head injury, or greater than or equal to 2 concussions within last year).
9. Current involvement in a weight loss program, participating in psychotherapy aimed at weight loss or treatment of eating behavior (e.g., binge eating).
10. All parents/guardians will be asked to indicate if their child has any food allergies. To be conservative, children who report allergies to gluten, nuts, dairy, fruit, or any other item in the array, will be excluded from the test meal portion of the study.
11. A condition under which MEG is contradicted (e.g., metal in the body, pregnancy, claustrophobia, history of significant neurological insult or injury).
12. Non-English speaking participants will be excluded from the study as they may be unable to complete questionnaires and follow the instructions which are only provided in English.

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: NIH subject data will become available starting 6 months after publication of a results paper and will be available from the NIH site for 2 years.
Access Criteria: NIH data with personal identifiers removed will be shared upon reasonable request to the PI, who will review requests. A data sharing agreement will be required to be negotiated with NICHD before sharing takes place.

REFERENCES:
- [Background] Shank LM, Tanofsky-Kraff M, Nelson EE, Shomaker LB, Ranzenhofer LM, Hannallah LM, Field SE, Vannucci A, Bongiorno DM, Brady SM, Condarco T, Demidowich A, Kelly NR, Cassidy O, Simmons WK, Engel SG, Pine DS, Yanovski JA. Attentional bias to food cues in youth with loss of control eating. Appetite. 2015 Apr;87:68-75. doi: 10.1016/j.appet.2014.11.027. Epub 2014 Nov 27. PMID 25435490
- [Background] Waters AM, Lipp OV, Spence SH. Attentional bias toward fear-related stimuli: an investigation with nonselected children and adults and children with anxiety disorders. J Exp Child Psychol. 2004 Dec;89(4):320-37. doi: 10.1016/j.jecp.2004.06.003. PMID 15560877
- [Background] Jarcho JM, Tanofsky-Kraff M, Nelson EE, Engel SG, Vannucci A, Field SE, Romer AL, Hannallah L, Brady SM, Demidowich AP, Shomaker LB, Courville AB, Pine DS, Yanovski JA. Neural activation during anticipated peer evaluation and laboratory meal intake in overweight girls with and without loss of control eating. Neuroimage. 2015 Mar;108:343-53. doi: 10.1016/j.neuroimage.2014.12.054. Epub 2014 Dec 27. PMID 25550068
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-CH-0014.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2/10/2017 to 4/27/2023 from the local community by advertisements sent by mail and posted flyers.
Groups:
- AB Control: Control condition - the probe is equally likely to replace the food picture and the neutral picture. There is no correlation between picture type and probe location, and no training of attention should occur.
  Attention Bias Retraining: Attention retraining program on smartphone where the probe always replaces the neutral picture. There is a perfect correlation between picture type and probe location.
Period: Overall Study
Arm/Group | AB Control | AB Retraining
Started | 36 | 32
Completed | 29 | 29
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Population: 68 were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | AB Control | AB Retraining | Total
Number analyzed (Participants) | 36 | 32 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (1.7) | 15.0 (1.6) | 14.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 68
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 18 | 37
  White | 14 | 8 | 22
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 36 | 32 | 68
Fat Mass [Mean (Standard Deviation); unit: Kg] — Fat mass, measured by dual-energy x-ray absorptiometry iDXA, Lunar.
  Kg | 33.6 (11.3) | 33.8 (10.4) | 33.7 (10.8)
Body Mass Index Z-score [Mean (Standard Deviation); unit: Z-score] — Body Mass Index (BMI) Z-score for age and sex, calculated according to the US Centers for Disease Control recommended approach. Z-scores represent the number of standard deviations of a value from the mean. BMI Z-scores of 0 represent the mean BMI for sex and age, above 0 represent above-average BMI for sex and age, and below 0 represent below-average BMI for sex and age. A BMI Z-score between 1.04 and 1.64 indicates overweight. A BMI Z-score greater than 1.64 indicates obesity.
  Z-score | 1.88 (0.64) | 1.80 (0.55) | 1.84 (0.60)
Recent Loss Of Control Eating [Count of Participants; unit: Participants] — Determined through the Eating Disorder Examination semi-structured interview. Number of participants reporting loss of control over their eating within the past 1 month.
  Participants | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Changes in Food-cue Visual Probe Task Attention Bias (AB) Reaction Time
Description: AB was obtained for each stimulus pairing (High-Palatability Food [HPF] minus Non-Food [NF] image, Low-Palatability Food [LPF] minus NF image, HPF minus LPF image). Trials where the probe appeared behind the more food-salient cue (e.g., a HPF image, or LPF vs NF image) were considered congruent trials. Trials where the probe appeared behind the less salient cue (e.g., NF image, or LPF image when the other image was a HPF image) were considered incongruent trials. The average reaction time during incongruent trials was subtracted from reaction time during during congruent trials. Positive scores represent a quicker reaction time for (and bias towards) the more palatable stimulus, and negative scores represent a slower reaction time for (and bias away from) the more palatable stimulus. A difference score of 0 represents no bias towards or away from the more palatable stimulus. Only trials with correct responses for the direction of the probe were included in computations.
Time Frame: 2-weeks
Population: Computer failures led to missing data for many participants. There were interruptions in data recording during magnetoencephalography sessions that were not predictable due to equipment failures.
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in milliseconds
Arm/Group | AB Retraining | Control Sham
Number analyzed (Participants) | 22 | 21
Change in milliseconds | 1.85 [-8.44 to 12.13] | 4.27 [-6.25 to 14.80]
Statistical Analysis 1: Comparison: AB Retraining vs Control Sham; Sample size estimation was based on the power analysis for the first hypothesis (examine changes in AB following completion of the smartphone program). Assuming 35% attrition, 80 girls, 40 with LOC-eating and 40 without LOC-eating, were estimated to provide >80% power to detect medium to large effects; Test type: Superiority — Change scores were computed (post-intervention - pre-intervention = delta) for AB reaction time measures. A linear mixed model was run with change scores as the dependent variable. Between-subject factors were condition, recent LOC-eating (0=absent, 1=present), and a condition by LOC-eating interaction term. AB reaction times were nested within subject. Models included a random intercept and were adjusted for stimuli pairing type, age, fat mass, height, and race and ethnicity; Effect sizes and 95% CIs, rather than statistical significance, were used. Cohen's d was interpreted as minimal to no effect (<.02) small effect (0.2-0.49) medium effect (0.5-0.79) large effect (0.8); beta coefficient = -1.948, 95% CI 2-sided [-20.790 to 16.894] — To examine changes in AB, change scores were computed (post-pre = delta). Positive scores represent an increase in AB from pre- to post- intervention. Negative ∆reaction time scores represent a decrease in AB from pre- to post- intervention
Statistical Analysis 2: Comparison: AB Retraining vs Control Sham; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.952, 95% CI 2-sided [-35.280 to 33.377]

2. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudate Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power at the caudate left hemisphere during attention capture (0-250ms following stimulus). Oscillatory power was normalized as per NeuroImage 39 (2008) pp 1788-1802, by estimating noise power as ρθ = WθTΣWθ (where Wθ is a (M × 1) column vector of weighting parameters that are tuned specifically to the location and orientation represented by θ, Σ represents the noise covariance matrix and ρθ is the beamformer-projected sensor noise power at the location and orientation θ). Within each stimuli-pairing and attention phase, oscillatory power during the incongruent trials was divided by oscillatory power during the congruent trials, then log transformed. Given a ratio was used, the oscillator power outcomes are unitless. Change in power (post-intervention minus pre-intervention) was calculated. Positive changes represent an increase in oscillatory power from pre- to post intervention.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.010 [-0.027 to 0.048] | .021 [-0.014 to 0.056]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; Sample size estimation was based on the power analysis for the first hypothesis (examine changes in oscillatory power following completion of the smartphone program). Assuming 35% attrition, 80 girls, 40 with LOC-eating and 40 without LOC-eating, were estimated to provide >80% power to detect medium to large effects; Test type: Superiority — Change scores were computed (post-intervention - pre-intervention = delta) for oscillatory power. A linear mixed model was run with change scores as the dependent variable. Between-subject factors were condition, recent LOC-eating (0=absent, 1=present), and a condition by LOC-eating interaction term. Oscillatory power analyses were nested within subject. Models included a random intercept and were adjusted for stimuli pairing type, age, fat mass, height, and race and ethnicity; [p-value comment as in outcome 1, analysis 1]; beta coefficent = 0.047, 95% CI 2-sided [-0.025 to 0.119] — To examine changes in oscillatory power, change scores were computed (post-pre=delta). Positive scores represent an increase from pre- to post- intervention. Negative scores represent a decrease from pre- to post- intervention
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.134, 95% CI 2-sided [-0.288 to 0.019]

3. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudate Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the caudate right hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.032 [-0.011 to 0.075] | 0.023 [-0.017 to 0.063]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Change scores were computed (post-intervention - pre-intervention = delta) for oscillatory power. A linear mixed model was run with change scores as the dependent variable. Between-subject factors were condition, recent LOC-eating (0=absent, 1=present), and a condition by LOC-eating interaction term. Oscillatory power analyses were nested within subject. Models included a random intercept and were adjusted for stimuli pairing type, age, fat mass and height, race and ethnicity; [p-value comment as in outcome 1, analysis 1]; beta coefficent = -0.002, 95% CI 2-sided [-0.085 to 0.082] — To examine changes in oscillatory power, change scores were computed (post-pre=delta). Positive scores represent an increase from pre- to post-intervention. Negative scores represent a decrease from pre- to post- intervention
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.053, 95% CI 2-sided [-0.177 to 0.071]

4. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pallidum Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pallidum left hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.007 [-0.055 to 0.041] | 0.038 [-0.006 to 0.083]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.080, 95% CI 2-sided [-0.022 to 0.182] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.018, 95% CI 2-sided [-0.139 to 0.103]

5. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pallidum Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pallidum right hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.028 [-0.022 to 0.078] | 0.009 [-0.037 to 0.056]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.013, 95% CI 2-sided [-0.086 to 0.113] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.035, 95% CI 2-sided [-0.179 to 0.109]

6. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Putamen Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the putamen left hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.013 [-0.056 to 0.030] | 0.046 [0.006 to 0.086]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.083, 95% CI 2-sided [-0.001 to 0.167] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.069, 95% CI 2-sided [-0.201 to 0.063]

7. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Putamen Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the putamen right hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.017 [-0.029 to 0.063] | 0.020 [-0.022 to 0.063]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.031, 95% CI 2-sided [-0.059 to 0.121] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.002, 95% CI 2-sided [-0.157 to 0.152]

8. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudal Anterior Cingulate Cortex Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the caudal anterior cingulate cortex left hemisphere - during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.035 [-0.009 to 0.078] | -0.041 [-0.081 to -0.001]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.042, 95% CI 2-sided [-0.149 to 0.065] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.068, 95% CI 2-sided [-0.266 to 0.131]

9. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudal Anterior Cingulate Cortex Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the caudal anterior cingulate cortex right hemisphere - during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.053 [0.011 to 0.095] | 0.002 [-0.037 to 0.041]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.034, 95% CI 2-sided [-0.122 to 0.053] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.070, 95% CI 2-sided [-0.233 to 0.092]

10. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Rostral Anterior Cingulate Cortex Left Hemisphere - During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the rostral anterior cingulate cortex left hemisphere - during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.012 [-0.030 to 0.055] | 0.012 [-0.027 to 0.051]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.042, 95% CI 2-sided [-0.041 to 0.126] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.085, 95% CI 2-sided [-0.252 to 0.082]

11. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Rostral Anterior Cingulate Cortex Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the rostral anterior cingulate cortex right hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.002 [-0.034 to 0.039] | -0.024 [-0.058 to 0.010]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.021, 95% CI 2-sided [-0.060 to 0.102] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.071, 95% CI 2-sided [-0.260 to 0.119]

12. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Lateral Orbitofrontal Cortex Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Neural activity during a food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the lateral orbitofrontal cortex left hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.010 [-0.050 to 0.030] | 0.026 [-0.011 to 0.063]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.107, 95% CI 2-sided [0.030 to 0.185] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.197, 95% CI 2-sided [-0.346 to -0.047]

13. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Lateral Orbitofrontal Cortex Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the lateral orbitofrontal cortex right hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.026 [-0.065 to 0.014] | -0.001 [-0.037 to 0.036]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.092, 95% CI 2-sided [0.010 to 0.175] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.049, 95% CI 2-sided [-0.204 to 0.107]

14. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Medial Orbitofrontal Cortex Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the medial orbitofrontal cortex left hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.010 [-0.048 to 0.029] | 0.018 [-0.017 to 0.054]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.046, 95% CI 2-sided [-0.032 to 0.123] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = 0.007, 95% CI 2-sided [-0.163 to 0.177]

15. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Medial Orbitofrontal Cortex Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the medial orbitofrontal cortex right hemisphere during attention capture (0-250ms following stimulus).The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.018 [-0.053 to 0.018] | -0.011 [-0.044 to 0.022]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.041, 95% CI 2-sided [-0.03 to 0.112] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.014, 95% CI 2-sided [-0.168 to 0.140]

16. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudal Dorsolateral Prefrontal Cortex Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the caudal dorsolateral prefrontal cortex left hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.026 [-0.006 to 0.058] | 0.020 [-0.010 to 0.049]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.037, 95% CI 2-sided [-0.125 to 0.052] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.034, 95% CI 2-sided [-0.196 to 0.129]

17. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudal Dorsolateral Prefrontal Cortex Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the caudal dorsolateral prefrontal cortex right hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.027 [-0.010 to 0.065] | 0.031 [-0.003 to 0.066]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.001, 95% CI 2-sided [-0.091 to 0.093] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.143, 95% CI 2-sided [-0.286 to 0.001]

18. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Rostral Dorsolateral Prefrontal Cortex Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the rostral dorsolateral prefrontal cortex left hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.006 [-0.040 to 0.029] | 0.033 [0.001 to 0.066]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.065, 95% CI 2-sided [-0.001 to 0.132] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.095, 95% CI 2-sided [-0.246 to 0.055]

19. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Rostral Dorsolateral Prefrontal Cortex Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the rostral dorsolateral prefrontal cortex right hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.014 [-0.018 to 0.046] | 0.008 [-0.021 to 0.038]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.023, 95% CI 2-sided [-0.055 to 0.101] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.020, 95% CI 2-sided [-0.178 to 0.137]

20. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Superior Dorsolateral Prefrontal Cortex Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the superior dorsolateral prefrontal cortex left hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.021 [-0.004 to 0.046] | -0.013 [-0.036 to 0.010]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.032, 95% CI 2-sided [-0.116 to 0.051] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = 0.060, 95% CI 2-sided [-0.104 to 0.223]

21. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Superior Dorsolateral Prefrontal Cortex Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the superior dorsolateral prefrontal cortex right hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.041 [0.017 to 0.064] | 0.019 [-0.002 to 0.041]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.012, 95% CI 2-sided [-0.078 to 0.053] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.064, 95% CI 2-sided [-0.248 to 0.120]

22. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Opercularis Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars opercularis left hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.010 [-0.048 to 0.029] | 0.069 [0.034 to 0.105]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.089, 95% CI 2-sided [0.004 to 0.174] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = 0.021, 95% CI 2-sided [-0.159 to 0.201]

23. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Opercularis Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars opercularis right hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.037 [-0.007 to 0.080] | 0.031 [-0.009 to 0.071]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.016, 95% CI 2-sided [-0.113 to 0.081] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.072, 95% CI 2-sided [-0.206 to 0.062]

24. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Orbitalis Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars orbitalis left hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.019 [-0.060 to 0.023] | 0.019 [-0.019 to 0.058]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.129, 95% CI 2-sided [0.049 to 0.209] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.181, 95% CI 2-sided [-0.330 to -0.033]

25. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Orbitalis Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars orbitalis right hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.011 [-0.053 to 0.030] | 0.016 [-0.023 to 0.055]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.126, 95% CI 2-sided [0.045 to 0.207] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.056, 95% CI 2-sided [-0.223 to 0.112]

26. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Triangularis Left Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars triangularis left hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.015 [-0.059 to 0.029] | 0.064 [0.024 to 0.105]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.115, 95% CI 2-sided [0.027 to 0.203] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.058, 95% CI 2-sided [-0.203 to 0.087]

27. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Triangularis Right Hemisphere During Attention Capture (0-250ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars triangularis right hemisphere during attention capture (0-250ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.022 [-0.020 to 0.063] | 0.016 [-0.023 to 0.054]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.037, 95% CI 2-sided [-0.053 to 0.127] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.085, 95% CI 2-sided [-0.240 to 0.069]

28. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudate Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the the caudate left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.012 [-0.025 to 0.049] | -0.052 [-0.086 to -0.017]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.021, 95% CI 2-sided [-0.092 to 0.050] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.096, 95% CI 2-sided [-0.249 to 0.056]

29. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudate Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the caudate right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.030 [-0.013 to 0.073] | -0.031 [-0.070 to 0.009]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.013, 95% CI 2-sided [-0.095 to 0.069] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.078, 95% CI 2-sided [-0.227 to 0.071]

30. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pallidum Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pallidum left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.011 [-0.058 to 0.036] | -0.051 [-0.095 to -0.008]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.005, 95% CI 2-sided [-0.103 to 0.092] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.032, 95% CI 2-sided [-0.173 to 0.110]

31. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pallidum Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pallidum right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.037 [-0.009 to 0.084] | -0.026 [-0.069 to 0.017]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.020, 95% CI 2-sided [-0.069 to 0.109] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.088, 95% CI 2-sided [-0.252 to 0.077]

32. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Putamen Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the putamen left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.0005 [-0.040 to 0.041] | -0.062 [-0.100 to -0.025]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.010, 95% CI 2-sided [-0.099 to 0.080] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.155, 95% CI 2-sided [-0.294 to -0.017]

33. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Putamen Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the putamen right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.018 [-0.024 to 0.061] | -0.031 [-0.070 to 0.009]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.013, 95% CI 2-sided [-0.069 to 0.095] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.085, 95% CI 2-sided [-0.216 to 0.047]

34. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudal Anterior Cingulate Cortex Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the caudal anterior cingulate cortex left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.026 [-0.012 to 0.064] | -0.069 [-0.104 to -0.033]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.041, 95% CI 2-sided [-0.123 to 0.041] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.096, 95% CI 2-sided [-0.213 to 0.021]

35. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudal Anterior Cingulate Cortex Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the caudal anterior cingulate cortex right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.058 [0.011 to 0.105] | -0.028 [-0.072 to 0.016]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.038, 95% CI 2-sided [-0.142 to 0.066] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.096, 95% CI 2-sided [-0.290 to 0.097]

36. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Rostral Anterior Cingulate Cortex Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the rostral anterior cingulate cortex left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.005 [-0.048 to 0.038] | -0.030 [-0.070 to 0.010]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.023, 95% CI 2-sided [-0.105 to 0.059] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.124, 95% CI 2-sided [-0.277 to 0.029]

37. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Rostral Anterior Cingulate Cortex Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the rostral anterior cingulate cortex right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.032 [-0.010 to 0.074] | -0.012 [-0.051 to 0.027]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.057, 95% CI 2-sided [-0.140 to 0.027] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.161, 95% CI 2-sided [-0.302 to -0.020]

38. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Lateral Orbitofrontal Cortex Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the lateral orbitofrontal cortex left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.021 [-0.022 to 0.063] | -0.062 [-0.102 to -0.023]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.0002, 95% CI 2-sided [-0.091 to 0.091] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.004, 95% CI 2-sided [-0.157 to 0.149]

39. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Lateral Orbitofrontal Cortex Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the lateral orbitofrontal cortex right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.012 [-0.029 to 0.052] | 0.002 [-0.035 to 0.040]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.010, 95% CI 2-sided [-0.092 to 0.071] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = 0.029, 95% CI 2-sided [-0.126 to 0.183]

40. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Medial Orbitofrontal Cortex Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the medial orbitofrontal cortex left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.018 [-0.023 to 0.058] | -0.038 [-0.076 to -0.001]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.013, 95% CI 2-sided [-0.101 to 0.076] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.106, 95% CI 2-sided [-0.273 to 0.060]

41. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Medial Orbitofrontal Cortex Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the medial orbitofrontal cortex right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.041 [0.001 to 0.080] | -0.009 [-0.046 to 0.028]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.033, 95% CI 2-sided [-0.110 to 0.043] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.166, 95% CI 2-sided [-0.335 to 0.003]

42. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudal Dorsolateral Prefrontal Cortex Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the caudal dorsolateral prefrontal cortex left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.016 [-0.024 to 0.056] | -0.012 [-0.049 to 0.025]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.011, 95% CI 2-sided [-0.069 to 0.091] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.167, 95% CI 2-sided [-0.332 to -0.002]

43. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Caudal Dorsolateral Prefrontal Cortex Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the caudal dorsolateral prefrontal cortex right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.005 [-0.041 to 0.050] | 0.006 [-0.036 to 0.048]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.054, 95% CI 2-sided [-0.037 to 0.146] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.019, 95% CI 2-sided [-0.127 to 0.090]

44. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Rostral Dorsolateral Prefrontal Cortex Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the rostral dorsolateral prefrontal cortex left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.015 [-0.017 to 0.047] | -0.031 [-0.061 to -0.002]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.002, 95% CI 2-sided [-0.061 to 0.065] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.086, 95% CI 2-sided [-0.215 to 0.042]

45. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Rostral Dorsolateral Prefrontal Cortex Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the rostral dorsolateral prefrontal cortex right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.010 [-0.024 to 0.044] | -0.006 [-0.037 to 0.026]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.032, 95% CI 2-sided [-0.05 to 0.115] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.095, 95% CI 2-sided [-0.248 to 0.058]

46. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Superior Dorsolateral Prefrontal Cortex Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the superior dorsolateral prefrontal cortex left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.004 [-0.025 to 0.033] | -0.022 [-0.049 to 0.005]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.016, 95% CI 2-sided [-0.075 to 0.042] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = 0.025, 95% CI 2-sided [-0.130 to 0.180]

47. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Superior Dorsolateral Prefrontal Cortex Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the superior dorsolateral prefrontal cortex right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.023 [-0.009 to 0.055] | 0.010 [-0.020 to 0.039]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.030, 95% CI 2-sided [-0.039 to 0.099]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.143, 95% CI 2-sided [-0.335 to 0.049]

48. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Opercularis Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars opercularis left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.043 [0.003 to 0.082] | -0.054 [-0.09 to -0.017]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.016, 95% CI 2-sided [-0.097 to 0.066] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.162, 95% CI 2-sided [-0.314 to -0.01]

49. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Opercularis Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars opercularis right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.001 [-0.037 to 0.039] | -0.018 [-0.053 to 0.017]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.053, 95% CI 2-sided [-0.051 to 0.156] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.070, 95% CI 2-sided [-0.251 to 0.111]

50. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Orbitalis Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars orbitalis left hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.013 [-0.026 to 0.053] | -0.052 [-0.089 to -0.016]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.015, 95% CI 2-sided [-0.061 to 0.091] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.108, 95% CI 2-sided [-0.260 to 0.044]

51. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Orbitalis Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars orbitalis right hemisphere during attention deployment (250-500ms following stimulus).The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.027 [-0.067 to 0.012] | 0.023 [-0.014 to 0.060]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.036, 95% CI 2-sided [-0.047 to 0.119] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.106, 95% CI 2-sided [-0.276 to 0.064]

52. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Triangularis Left Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars triangularis left hemisphere during attention deployment (250-500ms following stimulus).The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | 0.023 [-0.015 to 0.062] | -0.071 [-0.107 to -0.036]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = -0.017, 95% CI 2-sided [-0.092 to 0.057] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = 0.002, 95% CI 2-sided [-0.150 to 0.153]

53. Primary Outcome: Change in Beta Band (13-35 Hz) Oscillatory Power During Food-cue Visual Probe Attention Bias Task in the Pars Triangularis Right Hemisphere During Attention Deployment (250-500ms Following Stimulus)
Description: Change in beta band (13-35 Hz) oscillatory power during food-cue visual probe attention bias task completed at the baseline laboratory visit vs. post-EMA intervention visit (conducted 2 weeks after the baseline visit) at the pars triangularis right hemisphere during attention deployment (250-500ms following stimulus). The same analysis procedure was followed as described in detail for the first primary outcome.
Time Frame: 2-weeks
Population: Equipment failure meant many participants did not have data for this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless
Arm/Group | AB Control | AB Retraining
Number analyzed (Participants) | 12 | 14
unitless | -0.009 [-0.055 to 0.037] | 0.013 [-0.030 to 0.056]
Statistical Analysis 1: Comparison: AB Control vs AB Retraining; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; [p-value comment as in outcome 1, analysis 1]; beta coefficient = 0.070, 95% CI 2-sided [-0.019 to 0.159] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AB Control vs AB Retraining; Interaction of Loss of Control Eating with attention bias. See Statistical Analysis 1 for details; Test type: Superiority — See Statistical Analysis 1 for details. No p-values supplied, only confidence intervals and Cohen's d; beta coefficient = -0.095, 95% CI 2-sided [-0.260 to 0.070]

54. Secondary Outcome: Frequency of Loss-of-control Eating Episodes
Description: Frequency of self-reported loss-of-control eating episodes measured via the Eating Disorder Examination Interview at the baseline visit and post-EMA intervention visit (conducted 2 weeks after the baseline visit).
Time Frame: 2-weeks
Population: Some subjects withdrew before completion of the post-smartphone visit.
Measure: Mean (Standard Deviation); unit: eating episode (count)
Arm/Group | AB Retraining | Control Sham
Number analyzed (Participants) | 26 | 26
eating episode (count) | .731 (2.3189) | .827 (1.968)
Statistical Analysis 1: Comparison: AB Retraining vs Control Sham; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.256, Generalized estimation equations; beta coefficient = -0.8707, Standard Error of Mean 0.766 — Reported variable is a condition by time (pre or post-intervention) interaction term. The model included a Poisson distribution, log link function, exchangeable covariance matrix and was adjusted for age, fat mass, height, and race and ethnicity

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | AB Retraining | Control Sham
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/36
Other Adverse Events (participants affected / at risk) | 4/32 | 2/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB Retraining (N=32) | Control Sham (N=36)
Headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Grade 1, During magnetoencephalography. MedDRA 10019211
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) — Grade 1, MedDRA 10028813
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 1, MedDRA 10028836

LIMITATIONS AND CAVEATS:
The primary study limitation was the small sample size and difficulties with recruitment. Other limitations include a large percentage of missing MEG data. Girls who provided complete data were, on average, older than participants who had missing data. Lastly, visual probe tasks have been shown to have relatively poor psychometric reliability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT02977403/Prot_SAP_000.pdf